CLINICAL TRIAL: NCT04954768
Title: Epidemiological Characteristics of Elderly Trauma Patients in Zhejiang Province and Development of Geriatric Trauma Short-term Mortality Prediction Model
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-038
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Trauma Injury; Old Injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — This is a observational study, and there is no interventions.

SUMMARY:
This is a retrospective study. Trauma patients aged 65 years or older will be included. The aims of this study are explore the epidemiological characteristics of elderly trauma patients in Zhejiang Province; establishment of early warning score system of elderly trauma death in Zhejiang Province; and horizontal comparison of the treatment level of elderly trauma in Zhejiang Province.

ELIGIBILITY:
Inclusion Criteria:

Trauma patients aged 65 years or older

Exclusion Criteria:

Secondary trauma due to other causes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Trauma patients aged 65 years or older
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
the incidence of geriatric trauma in patients | one year

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang university, school of medicine., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided